CLINICAL TRIAL: NCT05483231
Title: The Effect of Family Integrated Care on Melatonin Level in Very Low Birth Weight Infants in Neonatal Intensive Care Unit: A Multicenter Randomized Controlled Trial
Brief Title: The Effect of Family Integrated Care on Melatonin Level in Very Low Birth Weight Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-453
Record Dates: First submitted 2022-06-28; First posted 2022-08-02 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Very Low Birth Weight Infant
Keywords: Family integrated care; Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family integrated care intervention group (Experimental): Provide Family integrated care for very low birth weight infants in the NICU.
  Interventions: Behavioral: Family integrated care intervention group
- Routine nursing care group (Other): Perform routine nursing care for very low birth weight infants in the NICU.
  Interventions: Behavioral: Routine nursing care group

INTERVENTIONS:
Behavioral: Family integrated care intervention group — If the very low birth weight infants' vital signs are stable at 32 weeks of corrected gestational age, parents who have been fully trained will provide all non-medical care measures and developmental care for the VLBWIs in the NICU for not less than 6 hours per day for at least 3 weeks, and other medical practice and care measures will be the same as the routine group.
  Arms: Family integrated care intervention group
Behavioral: Routine nursing care group — Routine practice and in-hospital education will be given to the very low birth weight infants and parents. All care measures will be led by the nursing staff, without the participation of parents.
  Arms: Routine nursing care group

SUMMARY:
This study will explore the effect of Family integrated care (FICare) on the level of melatonin and other clinical outcomes in very low birth weight infants (VLBWIs) by integrating families into the neonatal intensive care unit (NICU) care team and participating in the daily care of VLBWIs, as well as the influence of FIcare on parents' outcomes.

DETAILED DESCRIPTION:
This study is a multicenter randomized controlled trial which mainly explores the effect of Family integrated care (FICare) on melatonin levels in very low birth weight infants (VLBWIs) in neonatal intensive care unit (NICU). The intervention group will use a FICare intervention program, mainly for families who have been fully trained by the NICU professional team and need to stay in the NICU to accompany and care for the VLBWIs for not less than 6 hours a day for at least 3 weeks. All non-medical care measures and developmental supportive care will be provided by parents as much as possible. The control group received routine nursing interventions in which all non-medical interventions are led by NICU staff and without parental involvement. The level of melatonin, clinical and parental outcomes in VLBWIs are compared between the intervention group and the control group to evaluate the effect of FICare intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1500g;
* Gestational age < 32w;
* Admit within 24 hours of birth;
* The parents are conscious and able to cooperate, have certain learning and reading comprehension skills, and are capable of caring for their babies. They are committed to receiving training and caring for their babies for not less than 6 hours a day for at least 21 days;
* Voluntarily participate in this study and sign informed consent.

Exclusion Criteria

* Newborns who require palliative care or surgical intervention;
* OI (oxygenation index) <300 ;
* Newborns with severe congenital malformations;

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes on the level of Melatonin in very low birth weight infants | From baseline to day 21 after the implementation of Family integrated care intervention
  At 32 weeks of corrected gestational age (baseline) and day 21 after the implementation of FICare intervention, melatonin will be quantitatively measured by high performance liquid chromatography-mass spectrometry (HPLC-MS) with saliva samples collected by a specially-assigned person.

SECONDARY OUTCOMES:
Breast feeding rate | At the day 21 after the implementation of Family integrated care intervention
  Data will be acquired at the day 21 after the implementation of FICare intervention by a specially-assigned person. Breastfeeding rate = number of VLBWI fed from mother's milk/total number of VLBWI enrolled in each group *100%.
Changes in maternal milk volume | From baseline to day 21 after the implementation of Family integrated care intervention
  At 32 weeks of corrected gestational age (baseline) and day 21 after the implementation of FICare intervention, maternal milk volume will be collected from lactation diary records issued before the intervention.
Rate of weight gain | From baseline to day 21 after the implementation of Family integrated care intervention
  Weight is measured by a parent or nurse. Rate of weight gain = ( Weight measured at day 21 after the intervention - weight measured at 32 weeks of corrected gestational age)/total number of intervention days.
Incidence of complications related to preterm birth | Through study completion, about an average of 21 days
  Complications related to preterm birth include neonatal sepsis, bronchopulmonary dysplasia (BPD), intraventicular hemorrhage (IVH), periventricular leukinomalacia (PVL), and retinopathy of prematurity (ROP). These complications are diagnosed by a neonatologist. If any of these conditions occurred during the intervention, complications related to preterm birth would be considered. Data will be obtained from the case system or data collection form.
Length of hospitalization | Through study completion, about an average of 21 days
  Length of hospitalization refers to the total number of days from 32 weeks of corrected gestational age (baseline) to the day of discharge. Data will be obtained from the case system.
Growth rate of head circumference | From baseline to day 21 after the implementation of Family integrated care intervention
  Head circumference is measured by a parent or nurse. Growth rate of head circumference = ( head circumference measured at day 21 after the intervention - head circumference measured at 32 weeks of corrected gestational age)/total number of intervention days.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Hu, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China